CLINICAL TRIAL: NCT04207112
Title: Economic Evaluation of New MDR TB Regimens (PRACTECAL EE)
Brief Title: Economic Evaluation of New MDR TB Regimens
Acronym: PRACTECAL-EE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Ministry of Health, Republic of Uzbekistan (Other Government); Ministry of Public Health, Republic of Belarus (Other Government); THINK TB & HIV Investigative Network (Network); University of Liverpool (Other); Wits Health Consortium (Pty) Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRACTECAL-EE
Record Dates: First submitted 2019-12-03; First posted 2019-12-20 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-01

CONDITIONS: Multi-drug Resistant Tuberculosis; Extensively Drug-Resistant Tuberculosis; Pulmonary Tuberculoses
Keywords: Bedaquiline; Pretomanid; Linezolid; Clofazimine; Moxifloxacin; Economic Evaluation; Pharmacoeconomics
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis, Pulmonary | interventions — bedaquiline; pretomanid; Moxifloxacin; Linezolid; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Moxifloxacin: 400 mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated Drug: Bedaquiline Bedaquiline is a diarylquinoline class antimicrobial which blocks the proton pump for ATP synthase of mycobacteria. This in turn blocks the ATP production required for cellular energy production and leading to cell death.
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Moxifloxacin; Drug: Linezolid
- Regimen 2: Bedaquiline, Pretomanid, Linezolid, Clofazimine (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated Clofazimine: 50 mg (less than 33 kg), 100 mg (more than 33 kg) for 24 weeks
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid; Drug: Clofazimine
- Regimen 3: Bedaquiline, Pretomanid, Linezolid (Experimental): Bedaquiline: 400 mg once daily for 2 weeks followed by 200 mg 3 times per week for 22 weeks Pretomanid: 200mg once daily for 24 weeks Linezolid: 600mg daily for 16 weeks then 300mg daily (or 600mg x3/wk) for the remaining 8 weeks or earlier when moderately tolerated)
  Interventions: Drug: Bedaquiline; Drug: Pretomanid; Drug: Linezolid
- Control regimen (Active Comparator): Locally accepted standard of care which is consistent with the WHO recommendations for the treatment of M/XDR-TB
  Interventions: Drug: Standard Drugs

INTERVENTIONS:
Drug: Bedaquiline — Bedaquiline is a diarylquinoline class antimicrobial which blocks the proton pump for ATP synthase of mycobacteria. This in turn blocks the ATP production required for cellular energy production and leading to cell death.
  Other Names: Sirturo; R207910; TMC207
  Arms: Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin; Regimen 2: Bedaquiline, Pretomanid, Linezolid, Clofazimine; Regimen 3: Bedaquiline, Pretomanid, Linezolid
Drug: Pretomanid — Pretomanid is an nitroimidazole class antimicrobial which interferes with cell wall biosynthesis in mycobacteria. It may have other mechanisms of action as well in non-replicating mycobacteria.
  Other Names: PA-824
  Arms: Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin; Regimen 2: Bedaquiline, Pretomanid, Linezolid, Clofazimine; Regimen 3: Bedaquiline, Pretomanid, Linezolid
Drug: Moxifloxacin — Moxifloxacin is an 8-methoxyquinolone class antimicrobial that is a potent inhibitor of DNA gyrase and topoisomerase IV in bacteria
  Other Names: Avelox; BAY 12-8039
  Arms: Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin
Drug: Linezolid — Linezolid, an oxazolidinone class antimicrobial which works by inhibiting ribosomal protein synthesis. It is approved for Gram-positive bacterial infections, and is increasingly being used for drug resistant TB disease.
  Other Names: Zyvox
  Arms: Regimen 1: Bedaquiline, Pretomanid, Linezolid, Moxifloxacin; Regimen 2: Bedaquiline, Pretomanid, Linezolid, Clofazimine; Regimen 3: Bedaquiline, Pretomanid, Linezolid
Drug: Clofazimine — Clofazimine (Cfz) is a lipophilic riminophenazine licensed for treatment of leprosy. Its mechanism(s) of action remains unclear, but existing evidence suggests production of reactive oxygen species within Mycobacterium tuberculosis is one mechanism.
  Other Names: Lamprene
  Arms: Regimen 2: Bedaquiline, Pretomanid, Linezolid, Clofazimine
Drug: Standard Drugs — Locally accepted standard of care which is consistent with the WHO recommendations for the treatment of M/XDR-TB.
  Arms: Control regimen

SUMMARY:
The current treatment regimen for MDR-TB has poor outcomes and costs of treating MDR-TB are greater than treating drug susceptible TB, both in terms of health service and patient-incurred costs. Urgent action is needed to Identify short, effective and tolerable treatments for people with MDR-TB. The PRACTECAL economic evaluation sub-study (PRACTECAL-EE) will take place alongside the TB PRACTECAL trial, aiming to assess the costs to patients and providers of such regimens and to estimate the cost-effectiveness and poverty impact of an introduction of new MDR-TB regimens in the three countries participating in the main study.

DETAILED DESCRIPTION:
Multidrug resistant tuberculosis (MDR TB), tuberculosis (TB) that does not respond to at least isoniazid and rifampicin, is currently a public health issue. The current treatment regimen for MDR-TB has poor outcomes and costs of treating MDR-TB are greater than treating drug susceptible TB, both in terms of health service and patient-incurred costs. (1, 2). Key changes to recommendations for MDR-TB treatment regimens were published recently by the World Health Organization after an assessment of new evidence(3). In this rapid communication, three main changes to the standard MDR regimen were recommended: firstly, the withdrawal of injectable antibiotics; secondly, the inclusion of bedaquiline in a recommended longer regimen (ie 20 months); and thirdly, the recommendation of use for a shorter regimen only for specific conditions. It also highlights the urgent need for evidence to inform better optimal treatment choices for MDR-TB patients. Economic evaluations of such bedaquiline-containing regimens will provide additional important information for decision makers who need to consider its economic value along with clinical efficacy when planning for introduction.

TB PRACTECAL is a randomised, controlled trial to evaluate the safety and efficacy of investigational regimens containing bedaquiline and pretomanid for the treatment of MDR-TB in adults. It has been designed in two stages: stage 1 is a phase II trial aiming to identify two regimens containing bedaquiline and pretomanid for further evaluation based on safety and efficacy outcomes after 8 weeks of treatment. Stage 2 is a phase III trial to evaluate the safety and efficacy of the two investigational regimens containing bedaquiline and pretomanid selected in stage 1 compared with the standard of care at 72 weeks post-randomisation (Clinical trial protocol, study number: NCT02589782). This economic evaluation sub-study (PRACTECAL EE) will take place alongside TB PRACTECAL aiming to assess the costs to patients and providers of such regimens and to estimate the cost-effectiveness and poverty impact of an introduction of new MDR-TB regimens in the three countries participating in the main study.

The decision problem is stated as the evaluation of the new treatment regimen for MDR TB patients to inform the GRADE process at a global level, and health technology assessments (HTA) in the trial host countries, as applied to regimens for drug-resistant TB. During these processes (both at global level, GRADE, and at country level, HTA), the review of economic evidence produced alongside clinical trials focuses around patient outcomes and then on resources needed to answer the question of whether a new regimen should be considered for introduction. Population level considerations can also be included, especially in a second stage where the decision problem has advanced from whether to recommend a new regimen, to how to introduce it to achieve maximum health at a limited budget.

The overall aim of this sub study is to estimate the probability that new MDR-TB regimens containing bedaquiline and pretomanid will be cost-effective from a societal as compared to the standard of care for MDR-TB patients in three settings: Uzbekistan, South Africa, and Belarus.

A secondary aim is to assess the costs from a provider perspective of treating patients with these new regimens (new MDR-TB regimens containing bedaquiline and pretomanid), and estimate the impact of new regimens on prevalence of catastrophic costs due to TB.

The specific objectives of this sub-study are, in each setting:

1. to assess the costs from a provider's perspective for selected facilities in the intervention and control arms;
2. to assess the costs from a patient's perspective for a sample of patients seeking care in study facilities in the intervention and control arms;
3. To estimate the prevalence of catastrophic costs in the intervention and control arms;
4. to assess the probability of new regimens being cost-effective at different willingness-to-pay thresholds from a societal perspective using a Markov model.

ELIGIBILITY:
Inclusion Criteria:

* adults with Mycobacterium tuberculosis resistant to at least rifampicin by either molecular or phenotypic drug susceptibility test.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Incremental cost incurred per disability adjusted life year (DALY) averted: Societal Perspective | 108 weeks post randomisation
  Incremental cost incurred per disability adjusted life year (DALY) averted with the intervention regimen compared to the standard of care from societal perspective. DALYs will be modelled up to a life time horizon using a markov model.
Incremental cost per disability adjusted life year (DALY) averted: Provider Perspective | 108 weeks post randomisation
  Incremental cost per disability adjusted life year (DALY) averted with the intervention regimen compared to the standard of care from provider perspective. DALYs will be modelled up to a life time horizon using a markov model.

SECONDARY OUTCOMES:
Mean cost per month of treatment | 108 weeks post randomisation
  Mean cost per month of treatment for different regimens and type of patient (MDR-TB, pre-XDR-TB (resistant to fluoroquinolone) and XDR-TB)
Mean cost per course of treatment for different types of patients | 108 weeks post randomisation
  Mean cost per course of treatment for different types of patients (MDR-TB, pre-XDR-TB (resistant to fluoroquinolone), XDR-TB) and by category (training, monitoring, service delivery and drugs)
Incremental total cost of intervention for the trial population | 108 weeks post randomisation
  Incremental total cost of intervention for the trial population, over the trial duration
Incremental total cost of intervention for the modelling cohort | 108 weeks post randomisation
  Incremental total cost of intervention for the modelling cohort, over a life time horizon

CONTACTS AND LOCATIONS:
Overall Officials: Sedona Sweeny, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (7):
- Republican Scientific and Practical Centre for Pulmonology and Tuberculosis hospital, Minsk, Belarus
- South Africa (4):
  - Helen Joseph Hospital, Johannesburg, Gauteng
  - THINK Clinical Trial Unit, Hillcrest, Durban, KwaZulu-Natal
  - King DinuZulu Hospital, Durban, KwaZulu-Natal
  - Doris Goodwin Hospital, Pietermaritzburg, KwaZulu-Natal
- Uzbekistan (2):
  - Republican TB Hospital No. 2, Nukus, Karakalpakstan
  - Sh Alimov Republican Specialised Scientific-Practical Medical Centre for Phthysiology and Pulmonology Hospital, Tashkent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweeney S, Gomez G, Kitson N, Sinha A, Yatskevich N, Staples S, Moodliar R, Motlhako S, Maloma M, Rassool M, Ngubane N, Ndlovu E, Nyang'wa BT. Cost-effectiveness of new MDR-TB regimens: study protocol for the TB-PRACTECAL economic evaluation substudy. BMJ Open. 2020 Oct 10;10(10):e036599. doi: 10.1136/bmjopen-2019-036599. PMID 33039989